CLINICAL TRIAL: NCT01103479
Title: Low-Literacy Physician-Patient Intervention Promoting Colorectal Cancer Screening
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Kenzie Cameron, Research Associate Professor, Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: R01CA140177-01 (NIH); R01CA140177 (NIH)
Record Dates: First submitted 2010-04-12; First posted 2010-04-14 (Estimated); Results first posted 2014-09-09 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Colorectal Cancer
Keywords: Early Detection of Cancer; Colorectal Cancer Screening
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Physicians

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Control (No Intervention): Participants will complete interviewer-administered pre- and post-test
- Physician Intervention (Experimental): Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer screening guidelines, communication skills, and health literacy training
  Interventions: Behavioral: Physician Intervention
- Physician and Patient Intervention (Experimental): Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer (CRC) screening guidelines, communication skills, and health literacy training; patients in this condition will also view an educational digital video disc (DVD) on CRC and CRC screening
  Interventions: Behavioral: Physician and Patient Intervention

INTERVENTIONS:
Behavioral: Physician Intervention — Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer (CRC) screening guidelines, communication skills, and health literacy training
  Arms: Physician Intervention
Behavioral: Physician and Patient Intervention — Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer (CRC) screening guidelines, communication skills, and health literacy training; patients in this condition will also view an educational DVD on CRC and CRC screening
  Arms: Physician and Patient Intervention

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a low literacy, physician and patient-directed intervention to promote colorectal cancer (CRC) screening among the medically underserved.

DETAILED DESCRIPTION:
This study will test the separate and combined effect of two of these interventions: 1) a provider communication skills training using a continuous quality improvement (CQI) framework, and 2) a brief, multimedia Patient Education Program (PEP) that incorporates plain language, graphic design, and audio voice-over to overcome literacy limitations. Our provider intervention has demonstrated efficacy to significantly improve CRC screening recommendation rates. Our multimedia program has also been field tested among patients with limited literacy and was able to improve patient knowledge and intention to receive screening.

We will implement both provider-only and combined provider-patient strategies within a federally qualified health center network to determine the most effective and efficient approach to promote CRC screening in these settings. Results from the study, supplemented by cost analyses and the process evaluation will directly inform translational strategies for cancer prevention within difficult community-based healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 50-75 years of age (in month 1 of the study)
* Patients have had two or more visits to the clinic during the past two years
* ACCESS Community Health Network patients
* University of Illinois Hospital & Health Sciences System patients
* Patients ages 50 - 75 as of the start of the intervention study
* English or Spanish-Speaking

Exclusion Criteria:

* Patients <50 or > 75 years of age
* Patients who have had fewer than two or more visits to the clinic during the past two years
* Personal history of CRC or colorectal polyps, or of inflammatory bowel disease and a family history with a first-degree relative with CRC or colorectal polyps.
* Unable to speak English or Spanish
* Compliant with CRC screening (FOBT or FIT within the past year; flexible sigmoidoscopy within past 5 years; colonoscopy within past 10 years)

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 569 (Actual)
Dates: Start 2010-04; Primary Completion 2013-07 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenzie A Cameron, PhD, Principal Investigator — Northwestern University
Locations (2):
- United States (2):
  - Access Community Health Network, Chicago, Illinois
  - University of Illinois Hospital & Health Sciences System, Chicago, Illinois

REFERENCES:
- [Derived] Cameron KA, Ramirez-Zohfeld V, Ferreira MR, Dolan NC, Radosta J, Galanter WL, Eder MM, Wolf MS, Rademaker AW. The Effects of a Multicomponent Colorectal Cancer Screening Intervention on Knowledge, Recommendation, and Screening among Underserved Populations. J Health Care Poor Underserved. 2020;31(4):1612-1633. doi: 10.1353/hpu.2020.0122. PMID 33416742
- [Derived] Ramirez-Zohfeld V, Rademaker AW, Dolan NC, Ferreira MR, Eder MM, Liu D, Wolf MS, Cameron KA. Comparing the Performance of the S-TOFHLA and NVS Among and Between English and Spanish Speakers. J Health Commun. 2015;20(12):1458-64. doi: 10.1080/10810730.2015.1018629. Epub 2015 Jul 6. PMID 26147770
- [Derived] Dolan NC, Ramirez-Zohfeld V, Rademaker AW, Ferreira MR, Galanter WL, Radosta J, Eder MM, Cameron KA. The Effectiveness of a Physician-Only and Physician-Patient Intervention on Colorectal Cancer Screening Discussions Between Providers and African American and Latino Patients. J Gen Intern Med. 2015 Dec;30(12):1780-7. doi: 10.1007/s11606-015-3381-8. Epub 2015 May 19. PMID 25986137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment for this study took place between September 15, 2010 and January 30, 2013 across seven federally qualified health centers as well as one large academic health center.
Pre-assignment Details: Enrolled participants were excluded from the trial before assignment to groups if they did not reach randomization (e.g. they did not reach the point in the pre-test survey where randomization took place. Therefore they were not assigned to groups. In this study, 3 of the 569 enrolled participants did not reach randomization.
Period: Overall Study
Arm/Group | Control | Physician Intervention | Physician and Patient Intervention
Started | 168 | 210 | 188
Completed | 163 | 201 | 174
Not Completed | 5 | 9 | 14
Not completed — Up to date with CRC screening | 1 | 9 | 12
Not completed — Family history of CRC | 1 | 0 | 2
Not completed — Active cancer | 1 | 0 | 0
Not completed — Saw non-study physician | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants had to reach randomization, complete both pre and post-tests, and be eligible for colorectal cancer screening (verified by chart review).
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Physician Intervention | Physician and Patient Intervention | Total
Number analyzed (Participants) | 163 | 201 | 174 | 538
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.46 (6.07) | 58.71 (6.24) | 57.03 (6.09) | 57.79 (6.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 124 | 144 | 129 | 397
  Male | 39 | 57 | 45 | 141
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic Black | 82 | 111 | 93 | 286
  Hispanic | 68 | 88 | 75 | 231
  Other/Missing | 13 | 2 | 6 | 21
Region of Enrollment [Number; unit: participants]
  United States | 163 | 201 | 174 | 538
Survey Language [Number; unit: participants]
  English | 100 | 118 | 106 | 324
  Spanish | 63 | 83 | 68 | 214
Insurance Status (more than one may apply) [Number; unit: participants]
  Private | 21 | 30 | 27 | 78
  Medicare | 47 | 68 | 52 | 167
  Medicaid | 51 | 71 | 67 | 189
  Uninsured | 66 | 52 | 42 | 160
Health Care System [Number; unit: participants]
  Community FQHC | 99 | 174 | 154 | 427
  Academic Health Center | 64 | 27 | 20 | 111
Years of Education [Number; unit: participants]
  0 - 6 years | 44 | 38 | 35 | 117
  7 - 12 years | 41 | 64 | 52 | 157
  13 or more years | 76 | 98 | 86 | 260
  Missing data | 2 | 1 | 1 | 4
Household Income [Number; unit: participants]
  <$20,000/year | 101 | 137 | 111 | 349
  $20,000 - $40,000/year | 22 | 28 | 23 | 73
  $40,001 - $100,000/year | 13 | 6 | 8 | 27
  Not sure/Don't know | 23 | 26 | 27 | 76
  Refused/Missing | 4 | 4 | 5 | 13
Health status [Number; unit: participants]
  Poor | 28 | 28 | 25 | 81
  Fair | 75 | 107 | 88 | 270
  Good | 39 | 46 | 44 | 129
  Very Good | 18 | 10 | 12 | 40
  Excellent | 2 | 10 | 4 | 16
  Missing | 1 | 0 | 1 | 2
Health Literacy [Number; unit: participants]
  Inadequate | 51 | 86 | 67 | 204
  Marginal/Adequate | 96 | 97 | 88 | 281
  Missing | 16 | 18 | 19 | 53

OUTCOME MEASURES:

1. Primary Outcome: Colorectal Cancer (CRC) Screening Completion
Description: CRC screening completion via Fecal Occult Blood Test (FOBT), Fecal Immunochemical Test (FIT) or Colonoscopy
Time Frame: within 6 months of provider recommendation
Measure: Number; unit: participants
Groups:
- Intervention: Participants in either the Physician Intervention or Physician and Patient Intervention Arms.
  Physician Intervention: Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer (CRC) screening guidelines, communication skills, and health literacy training
  Physician and Patient Intervention: Physician intervention as described plus patients in this condition will also view an educational digital video disc (DVD) on CRC and CRC screening
  Physician and Patient Intervention: Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer (CRC) screening guidelines, communication skills, and health literacy training; patients in this co
Arm/Group | Control | Intervention
Number analyzed (Participants) | 163 | 375
participants | 17 | 69
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.32, Mixed Models Analysis — Random effects model adjusting for clustering by clinic; Risk Ratio (RR) = 1.65, 95% CI 2-sided [0.62 to 4.38]

2. Primary Outcome: Colorectal Cancer (CRC) Screening Completion
Description: CRC screening completion via FOBT, FIT or Colonoscopy
Time Frame: within 6 months of provider recommendation
Measure: Number; unit: participants
Arm/Group | Physician Intervention | Physician and Patient Intervention
Number analyzed (Participants) | 201 | 174
participants | 41 | 28
Statistical Analysis 1: Comparison: Physician Intervention vs Physician and Patient Intervention; Test type: Superiority or Other; p = 0.28, Mixed Models Analysis — Linear model adjusting for stratification by clinic and participant age; Risk Ratio (RR) = 0.80, 95% CI 2-sided [0.53 to 1.20]

3. Secondary Outcome: Provider Recommendation of CRC Screening
Description: Provider recommendation of CRC Screening based on chart review
Time Frame: 6 months following patient enrollment into study
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 163 | 375
participants | 70 | 216
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority or Other; p = 0.42, Mixed Models Analysis — Random effects model adjusted for clustering by clinic; Risk Ratio (RR) = 1.43, 95% CI 2-sided [0.60 to 3.43]

4. Secondary Outcome: Provider Recommendation of CRC Screening
Description: Provider recommendation of CRC Screening based on chart review
Time Frame: 6 months following patient enrollment into study
Measure: Number; unit: participants
Arm/Group | Physician Intervention | Physician and Patient Intervention
Number analyzed (Participants) | 201 | 174
participants | 113 | 103
Statistical Analysis 1: Comparison: Physician Intervention vs Physician and Patient Intervention; Test type: Superiority or Other; p = 0.38, Mixed Models Analysis — Linear model adjusting for stratification by clinic and participant age; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.94 to 1.18]

ADVERSE EVENTS:
Groups:
- Physician Training: Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer screening guidelines, communication skills, and health literacy training
  Physician Intervention: Physicians at these clinics will participate in 6 training sessions over the course of 3 1/2 years; training sessions relate to colorectal cancer (CRC) screening guidelines, communication skills, and health literacy training
Arm/Group | Control | Physician Training | Physician and Patient Intervention
Serious Adverse Events (participants affected / at risk) | 0/163 | 0/201 | 0/174
Other Adverse Events (participants affected / at risk) | 0/163 | 0/201 | 0/174

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No